CLINICAL TRIAL: NCT06468085
Title: Clinical and Radiographic Evaluation of Premixed Bioceramic Putty and Biodentine™ Pulpotomy in Mature Permanent Anterior Teeth With Signs of Pulpitis: A Randomized Controlled Trial
Brief Title: Evaluation of Pulpotomy Using Two Different Agents in Mature Anterior Teeth With Pulpitis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Sally Emad Nathan Ghobrial, Assistant Lecturer, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FDASU-Rec ID032421
Record Dates: First submitted 2024-06-15; First posted 2024-06-21 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Pulpitis
MeSH Terms: conditions — Pulpitis | interventions — tricalcium silicate

STUDY DESIGN:
Intervention Model Description: two study groups and one control group
Who Masked: Participant
Masking Description: Double Blind study, where participants will be blinded to the study groups they are randomized to, statisticians will be blinded while performing statistical analysis. On the other hand, the operator/primary investigator cannot be blinded as she is already familiar with the tooth and materials used and their different application. Also, the outcome assessor is not blinded due to the difference between the used materials.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A: The premixed Bioceramic NeoPUTTY® group (Experimental): Cases will be evaluated clinically and radiographically to obtain baseline data. Local anesthesia will be administered and then rubber dam isolation will be performed. Pulpotomy procedure will be performed after hemostasis followed by covering pulp stump with Premixed Bioceramic NeoPUTTY® then final composite restoration will be applied.
  Interventions: Procedure: premixed Bioceramic NeoPUTTY®
- Group B: The Biodentine™ group (Experimental): Cases will be evaluated clinically and radiographically to obtain baseline data. Local anesthesia will be administered and then rubber dam isolation will be performed. Pulpotomy procedure will be performed after hemostasis followed by covering pulp stump with Biodentine™ then final composite restoration will be applied.
  Interventions: Procedure: Biodentine™
- Group C: the root canal treatment group (Active Comparator): Root canal treatment will be performed to the control group followed by composite restoration.
  Interventions: Procedure: Root canal treatment

INTERVENTIONS:
Procedure: premixed Bioceramic NeoPUTTY® — Pulpotomy procedure will be performed after hemostasis followed by covering pulp stump with Premixed Bioceramic then final composite restoration will be applied. clinical evaluation will be done at baseline, 3, 6, 9 and 12 months.
  Arms: Group A: The premixed Bioceramic NeoPUTTY® group
Procedure: Biodentine™ — Pulpotomy procedure will be performed after hemostasis followed by covering pulp stump with Premixed Bioceramic or Biodentine™ according to the corresponding group then final composite restoration will be applied. clinical evaluation will be done at baseline, 3, 6, 9 and 12 months.
  Arms: Group B: The Biodentine™ group
Procedure: Root canal treatment — Root canal treatment will be performed to the control group followed by composite restoration. clinical evaluation will be done at baseline, 3, 6, 9 and 12 months.
  Arms: Group C: the root canal treatment group

SUMMARY:
the study will evaluate the clinical and radiological success of mature permanent anterior teeth pulpotomy in children and adolescents with signs of pulpitis using two different Biomimetic materials (NeoPutty® and Biodentine™) as a pulp dressing material in comparison to root canal treatment at 3, 6, 9 and 12 months follow up.

DETAILED DESCRIPTION:
In this randomized controlled trial, A total number of 75 mature vital permanent anterior teeth with recent trauma or deep caries in children aged between 9 and 14 years will be included. Patients will be randomly allocated into three study groups: group A (premixed bioceramic NeoPutty®) test group, group B (Biodentine™) test group and group C (root canal treatment) control group. Cases will be evaluated clinically and radiographically to obtain baseline data. Local anesthesia will be administered and then rubber dam isolation will be performed. Pulpotomy procedure will be performed after hemostasis followed by covering pulp stump with Premixed Bioceramic or Biodentine™ according to the corresponding group then final composite restoration will be applied. Root canal treatment will be performed to the control group followed by composite restoration. Blinded clinical evaluation will be done at baseline, 3, 6, 9 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents of both sexes aged between 9 and 14 years old.
* Vital mature permanent anterior teeth with deep caries lesions that approach the pulp with signs of pulpitis and respond positive to cold pulp testing.
* Vital mature permanent anterior teeth with pulpal exposure that occurred during caries excavation.
* Patients presented immediately after suffering recent trauma (at the same day) to mature anterior teeth that had resulted in a crown fracture with pulp exposure.

Exclusion Criteria:

* Teeth with signs of infection such as swelling, sinus tract or pathological mobility or excessive mobility.
* Teeth with excessive bleeding from amputated radicular stumps
* Teeth showing radiographic evidence of pathologic root resorption, periapical pathology and calcifications in the canals.
* Lack of patient/parent compliance and cooperation.
* Children who are physically or mentally disabled or having any medical condition that will complicate the treatment.
* Patients allergic to any medicaments used.

Ages: 9 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 48 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Clinical success | 3, 6, 9 and 12 months follow up
  Absence of pain related to the treated teeth, including patient reported pain or sensitivity to percussion/palpation.
  No evidence of swelling of supporting soft tissue or presence of sinus tract. Absence of excessive mobility affecting treated teeth.
Radiographic success | 3, 6, 9 and 12 months follow up
  No Internal or external root resorption. No Periapical radiolucency.

SECONDARY OUTCOMES:
Evaluation of tooth discoloration. | 3, 6, 9 and 12 months follow up
  Evaluation of tooth discoloration using the VITA Easyshade V digital spectrophotometer.

CONTACTS AND LOCATIONS:
Overall Officials: Nagwa Khattab, BDS,MSc, MD, Study Director — Ain Shams University